CLINICAL TRIAL: NCT05165212
Title: Oral Amoxicillin Challenge in the Primary Care Setting
Brief Title: Primary Care Amoxicillin Challenge
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to host study at clinic site.
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Daniel Joseph Hamilton, Resident Physician, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00006018
Record Dates: First submitted 2021-12-20; First posted 2021-12-21 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Amoxicillin Allergy
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients receiving one dose of amoxicillin. (Experimental): Patients receiving one dose of amoxicillin and then observed for one hour for signs/symptoms off allergic reaction.
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — Patients will be given 10% of a standard weight-based dose of amoxicillin and observed for signs/symptoms of allergic reaction for 30 minutes. If no reaction occurs, they will given the remaining 90% of the standard dose and observed for an additional 30 minutes.

SUMMARY:
The purpose of this project is to identify clinic patients reporting penicillin allergy who are low risk for allergic reaction, and then invite them to participate in an oral amoxicillin challenge in their primary office without need for referral to allergy/immunology. If the patient is able to tolerate oral amoxicillin, the antibiotic allergy in question will be removed from the patient's chart.

DETAILED DESCRIPTION:
Patients with a documented allergy to amoxicillin, ampicillin, or penicillin who are deemed low-risk for true penicillin allergy based on history will be offered enrollment in the study. Patients will be scheduled for an oral amoxicillin challenge in the primary care office at a later date. During this challenge, patients will be given 10% of a weight-based dose of amoxicillin and then observed for 30 minutes for signs and symptoms of an allergic reaction. If no reaction occurs, they will be given the remaining 90% of the weight-based dose and observed for an additional 30 minutes. Emergency medications such as diphenhydramine and epinephrine will be immediately available if needed. If the patient completes oral amoxicillin challenge without a clinically significant reaction, penicillin (and/or amoxicillin/ampicillin) allergy will be removed from the patient's chart.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 18 years old who attend either of two hospital-affiliated general pediatric clinic sites who have an allergy to penicillin (or its derivatives) documented in their electronic medical record.

Exclusion Criteria:

* Patients who do not have an allergy to penicillin (or its derivatives) documented in their electronic medical record or patients with listed penicillin allergy whose parent/guardian declines to participate in the study. Patients will also be excluded if their penicillin allergy has been confirmed with either failed amoxicillin challenge or positive penicillin skin testing. Medically fragile children who cannot tolerate a direct oral challenge will be excluded but may be offered referral to allergy/immunology. If, on review of the history of the allergy, features of likely IgE mediated (onset in 1st hour of course or anaphylaxis requiring hospital care) or dangerous non-IgE mediated penicillin allergy (Stevens Johnson with penicillin, blistering rashes, penicillin related cytopenia) are obtained, these patients are also excluded from challenge but may be referred to allergy for further education and appropriate testing.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients reporting penicillin allergy | 12 months
  who are able to tolerate penicillin drug oral challenge in the primary care setting without prior referral to allergy/immunology.

IPD SHARING:
Plan to Share IPD: No